CLINICAL TRIAL: NCT06650592
Title: Objective Assessment of Outcomes Following Immediate Lymphatic Reconstruction / LYMPHA
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB24-1513
Record Dates: First submitted 2024-10-14; First posted 2024-10-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lymphatic Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients who were candidates for immediate lymphatic reconstruction (ILR): All patients who were candidates for immediate lymphatic reconstruction (ILR) in the LYMPHA Database
  Interventions: Other: All patients who were candidates for immediate lymphatic reconstruction (ILR)

INTERVENTIONS:
Other: All patients who were candidates for immediate lymphatic reconstruction (ILR) — All patients who were candidates for immediate lymphatic reconstruction (ILR)

SUMMARY:
Immediate lymphatic reconstruction (ILR) is a novel surgical approach performed at the time of initial lymph node dissection with the goal of preventing lymphedema. It involves the identification of lymphatic channels that are transected after lymph node dissection and microsurgical anastomosis of one or more lymphatic channel with a local recipient vein to re-direct upper extremity lymphatic drainage. Although ILR carries significant promise in prevention of lymphedema, there is a lack of high-level evidence supporting its efficacy because it is a novel surgical technique that is only offered at a few centers and not routinely covered by insurance carriers yet. The University of Chicago Comprehensive Cancer Center (UCCCC) is one of the busiest microsurgery centers performing this procedure, and, as a Lymphedema Center of Excellence, is in a unique position to investigate the efficacy of ILR in preventing lymphedema. In addition, the University has access to a world class microbiome research facility and colleagues. There is no information on the skin microbiome of the axilla in patients undergoing treatment for breast cancer or those at risk for developing lymphedema. Further exploratory studies such as this in a diverse patient population may lead to practice changing research in our approach to lymphedema management and prevention. The purpose of this study is to determine the role of immediate lymphatic reconstruction and obtain objective data to correlate the existing, self-reported rates of lymphedema at the University of Chicago.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were candidates for Immediate Lymphatic Reconstruction (ILR)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The University of Chicago has a prospectively maintained database (LYMPHA Database) of all patients who were candidates for ILR.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
The efficacy of immediate lymphatic reconstruction (ILR) based on objective circumference | 1 Day
the efficacy of immediate lymphatic reconstruction (ILR) based on volume | 1 Day
the efficacy of immediate lymphatic reconstruction (ILR) based on bioimpedance spectroscopy measurements of affected limbs of women in the prophylactic lymphedema database. | 1 Day
the efficacy of immediate lymphatic reconstruction (ILR) based on unaffected limbs of women in the prophylactic lymphedema database. | 1 Day

SECONDARY OUTCOMES:
the impact of ILR on validated patient reported outcome tool using the lymphedema life impact scale (LLIS) | 1 Day
  This is an 18 questionnaire that has a scale from 0 (no pain) to 4 (severe pain)
the impact of ILR on validated patient reported outcome tool using The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | 1 Day
  This is a 30 questionnaire that has a scale from 1 (No difficulty) to 5 (unable)
the impact of ILR on validated patient reported outcome tool using the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | 1 Day
  This is a 17 questionnaire that scales from unable to do it to not difficult.

OTHER OUTCOMES:
Axillary skin swabs of each axilla for microbiome analysis | 1 Day
  Characterize the axillary microbiome in limbs that have been treated with ILR compared to those that were unaffected.

CONTACTS AND LOCATIONS:
Overall Officials: Summer Hanson, MD, PhD, FACS, Principal Investigator — University of Chicago
Locations (1):
- The University o Chicago, Chicago, Illinois, United States